CLINICAL TRIAL: NCT04288466
Title: Gastric Emptying of Maltodextrin Solution in Elderly and in Adults: Clinical Trial
Brief Title: Gastric Emptying of Maltodextrin Solution in Elderly and in Adults
Acronym: GEMA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Brasilia University Hospital (Other)
Responsible Party: Principal Investigator, Gabriel Magalhaes Nunes Guimaraes, Clinical Professor, Brasilia University Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: tccandre2020
Record Dates: First submitted 2020-02-26; First posted 2020-02-28 (Actual); Last update posted 2020-02-28 (Actual); Status verified 2020-02

CONDITIONS: Aspiration; Liquids; Fasting; Perioperative Pulmonary Aspiration
MeSH Terms: conditions — Fasting | interventions — maltodextrin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Adults (Active Comparator): Adults < 60 years-old maltodextrin solution 450ml
  Interventions: Dietary Supplement: maltodextrin
- Elders (Active Comparator): Elders 65 or more years-old maltodextrin solution 450ml
  Interventions: Dietary Supplement: maltodextrin

INTERVENTIONS:
Dietary Supplement: maltodextrin — maltodextrin solution 450ml

SUMMARY:
Gastric volume will be measured before, 5, 30, 60, 90 and 120 min after drinking 450ml of maltodextrin in young adults and elderly.

DETAILED DESCRIPTION:
Gastric volume will be estimated before, 5, 30, 60, 90 and 120 min after drinking 450ml of maltodextrin in young adults and elderly using antral ultrasound.

ELIGIBILITY:
Inclusion Criteria:

* ASA physical status I or II;
* No known risk factor for slow or fast gastric emptying.

Exclusion Criteria:

* Vomiting the study solution before completion.
* Wrong timing of assessment.
* Protocol violation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2020-01-01 (Actual); Primary Completion 2020-04-01 (Estimated); Study Completion 2020-07-01 (Estimated)

PRIMARY OUTCOMES:
Antral Volume change | Just before and 5, 30, 60, 90 and 120 minutes after drinking the study solution (repeated measures)
  Antral volume in cm² assessed by ultrasound in semirecumbent position.

CONTACTS AND LOCATIONS:
Overall Officials: Gabriel MN Guimaraes, MSc, Principal Investigator — Professor
Locations (1):
- Hospital das Forças armadas, Brasília, Federal District, Brazil

IPD SHARING:
Plan to Share IPD: Yes
Plan to Share in Online Data Sharing Platform.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: We will put SAP and Analytic code in RPubs for as long as RPubs exists. Study protocol and ICF will be published in ClinicalTrials
Access Criteria: Open